CLINICAL TRIAL: NCT00529282
Title: Multicenter, Randomized, Double-Blind Study of Ceftobiprole Versus Comparators in the Treatment of Patients With Fever and Neutropenia
Brief Title: A Study of Ceftobiprole in Patients With Fever and Neutropenia.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued due to administrative reasons unrelated to safety
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014206; CEFTOFBN3004
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Results first posted 2010-03-29 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Fever; Neutropenia; Gram-positive Bacterial Infections; Pseudomonas Infection
Keywords: Low numbers of neutrophils in the blood; increased body temperature; cancer chemotherapy; ceftobiprole; pseudomonas infections
MeSH Terms: conditions — Fever; Neutropenia; Gram-Positive Bacterial Infections; Pseudomonas Infections | interventions — ceftobiprole medocaril; Cefepime; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Ceftobiprole Medocaril 500 mg every 8 hours 120-minute infusion [250 mL]
  Interventions: Drug: Ceftobiprole Medocaril
- 002 (Active Comparator): Cefepime with or without vancomycin 2 g every 8 hrs-30 min infusion vancomycin 1 000mg every 12 hrs-60 min infusion
  Interventions: Drug: Cefepime with or without vancomycin

INTERVENTIONS:
Drug: Ceftobiprole Medocaril — 500 mg every 8 hours
  Arms: 001
Drug: Cefepime with or without vancomycin — 120-minute infusion [250 mL]
  Arms: 002

SUMMARY:
The purpose of this study is to assess the safety and efficacy of ceftobiprole versus a comparator in patients with fever and neutropenia

DETAILED DESCRIPTION:
This study is being discontinued due to issues regarding the comparator, cefepime. In Nov 2007 FDA issued a MedWatch regarding cefepime and the trial was suspended. As of May 14, 2008 the FDA was still evaluating the data on cefepime and final follow up is pending. There were no safety issues with ceftobiprole in this study based on the enrollment of 2 subjects in September of 2007. The study is being discontinued for administrative reasons. Ceftobiprole medocaril is a cephalosporin antibiotic with anti-MRSA (Methicillin-Resistant Staphylococcus Aureus) activity. Ceftobiprole is not yet approved, but undergoing regulatory review for treatment of skin infections. This is a randomized (patients are assigned to receive the different treatments under study based on chance), double-blind (neither the patient nor the physician knows whether the drug being investigated or the comparator agent is being taken), multicenter study of treatment with ceftobiprole medocaril versus treatment with a comparator in patients 18 years of age or older, who have fever and neutropenia after chemotherapy for cancer that requires intravenous therapy. Patients will be randomly assigned to receive either ceftobiprole medocaril or comparator. In addition, patients in the comparator group who are at risk of serious infections due to gram-positive pathogens (disease-causing bacteria) may also receive an antibiotic with MRSA activity. The study will consist of the following 3 phases: a prerandomization phase (includes screening and baseline assessments); a treatment phase, and a follow-up phase consisting of a primary efficacy visit and a late follow-up visit. The primary endpoint is the clinical cure rate. The total duration of of the study is determined by the time to resolution of fever and neutropenia and the conditions associated with the episode of fever and neutropenia. This is followed by the primary efficacy visit (7 to 10 days after the end of therapy) and the late follow-up visit (28 to 35 days after the end of treatment). Cultures (samples of blood or other suspected sites of infection) will be collected during the study as well as blood samples for hematology and chemistry (safety assessments). All adverse events will also be reported throughout the study and for about 4 to 5 weeks after the last dose of study drug. Patients will be randomized to either ceftobiprole or comparator for approximately 7 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neutropenia and fever associated with administration of chemotherapy for cancer that requires intravenous therapy with antibiotics.

Exclusion Criteria:

* Patients who have received antibacterial (oral or intravenous ) treatment for more than 24 hours for fever and neutropenia or have received systemic antibacterial therapy in the previous 72 hours for a defined infectious disease
* Patients with known or suspected hypersensitivity to any related anti-infective
* patients with hepatic impairment
* Patients with severe renal impairment
* Patients who are pregnant or lactating
* Patients who are likely to require major surgical intervention for infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftobiprole Medocaril: 500 mg every 8 hours - 120-minute infusion [250 mL]
- Cefepime With or Without Vancomycin: 2 g every 8 hrs-30 min infusion vancomycin 1,000mg every 12 hrs-60 min infusion
Period: Overall Study
Arm/Group | Ceftobiprole Medocaril | Cefepime With or Without Vancomycin
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftobiprole Medocaril | Cefepime With or Without Vancomycin | Total
Number analyzed (Participants) | 0 | 2 | 2
Age Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 2 | 2
  >=65 years |  | 0 | 0
Gender [Number; unit: participants]
  Female |  | 1 | 1
  Male |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate of Ceftobiprole vs Comparator in Patients With Fever and Neutropenia.
Description: Clinical cure rate (the ratio of the number of clinically cured patients to the total number of patients in the population) at 7 to 10 days after end of therapy or before 24 hours of the initiation of the next course of chemotherapy, whichever is shorter. Cure without modification: A subject will be considered to be cured at the primary efficacy visit if: The subject's fever and clinical signs and symptoms are resolved to the extent that no further anti-infective therapy is necessary as determined by the investigator Any infecting organisms that were identified at baseline were eradicated
Time Frame: 7 to 10 days after end of therapy or before 24 hours of the initiation of the next course of chemotherapy, whichever is shorter.
Population: No outcome measures were analyzed due to early termination of the study.
Arm/Group | Ceftobiprole Medocaril | Cefepime With or Without Vancomycin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Clinical Cure Regardless of Modification of Therapy
Description: To demonstrate the noninferiority of ceftobiprole compared with cefepime with or without vancomycin with regard to clinical cure at the primary efficacy visit after completing the initial course of therapy, regardless of modification of therapy defined as addition of an anti-fungal agent and/or an aminoglycoside. Cure with modification: The subject requires antifungals, which will be considered a failure for the primary endpoint. The subject needs modification of study therapy by adding one or more agents (other than protocol-defined chemoprophylaxis antibiotics).
Time Frame: as for outcome 1
Population: No outcome measures were analyzed due to early termination of the study.
Arm/Group | Ceftobiprole Medocaril | Cefepime With or Without Vancomycin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Clinical Success at 72 Hours
Description: To compare the clinical success rate (absence or improvement of signs and symptoms of infection) at 72 hours after starting ceftobiprole with that of cefepime with or without vancomycin
Time Frame: 72 hours after starting study drug
Population: No outcome measures were analyzed due to early termination of the study.
Arm/Group | Ceftobiprole Medocaril | Cefepime With or Without Vancomycin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinical Cure Without Prophylactic Antibiotics After the End-of-treatment (EOT) Visit up to 28 Days of Study Drug
Description: To demonstrate the noninferiority of ceftobiprole compared with cefepime with or without vancomycin with regard to clinical cure at the primary efficacy visit after completing the unmodified initial course of therapy, and receiving no prophylactic antibiotics after the EOT visit.
Time Frame: as for outcome 1
Population: No outcome measures were analyzed due to early termination of the study.
Arm/Group | Ceftobiprole Medocaril | Cefepime With or Without Vancomycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The first subject completed on day 41 and the second subject completed on day 56.
Arm/Group | Ceftobiprole Medocaril | Cefepime With or Without Vancomycin
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/2
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftobiprole Medocaril (N=0) | Cefepime With or Without Vancomycin (N=2)
Bacteraemia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftobiprole Medocaril (N=0) | Cefepime With or Without Vancomycin (N=2)
Anorectal disorder (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
escherichia bacteremia (Infections and infestations) | 0 | 1
Catheter- related complication (General disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
No analysis was performed due to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days